CLINICAL TRIAL: NCT07286903
Title: Fluorescence Enhanced Stereotactic Surgery
Brief Title: Fluorescence Enhanced Stereotactic Surgery (FESS)
Acronym: FESS
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: FESS; PNRR-POC-2023-12377657 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: High Grade Glioma; High Grade Glioma (III or IV)
Keywords: Stereotactic Biopsy; Fluorescence Guided Surgery; 5-ALA; Raman Spectroscopy; Glioma; Fiber Opticts; Nashold Needle
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — standard IHC and molecular tests
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Histopathological diagnosis is essential for gliomas, but stereotactic biopsy carries significant risks and can fail to provide diagnostic tissue. This study aims to develop and validate an advanced fiber optic system integrated into a standard Nashold biopsy needle. This system combines 5-ALA fluorescence, Raman spectroscopy, and ultrasound imaging to provide real-time feedback on tumor tissue and blood vessels. The study involves ex-vivo testing on brain tumor tissues (High Grade Glioma) obtained through surgical resection to validate the system's ability to identify tumor margins and vascular structures, aiming to improve biopsy safety and accuracy.

DETAILED DESCRIPTION:
'The study focuses on the "Fluorescence Enhanced Stereotactic Surgery" (FESS) project. It is a prospective, multicenter, observational study on a device. The study consists of three phases:

Phase 1: Development and prototyping of fiber optic probes (by partner CERICT), integration into a standard biopsy needle, and software development.

Phase 2: In vitro testing on phantoms and ex-vivo testing on biological tissue. Ex-vivo tests will be performed on intra-axial brain tumor samples resected during standard surgery (guided by 5-ALA fluorescence). The probe will be inserted into the resected sample to detect fluorescence and vascular signals. Results will be correlated with histopathological analysis.

Phase 3: Optimization and final validation of the integrated system. Approximately 20 samples of high-grade glioma will be analyzed. The goal is to verify if the probe can distinguish tumor tissue (via 5-ALA fluorescence) and identify blood vessels (via ultrasound/Raman) to prevent hemorrhage during biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patients able to provide the informed consentPresumptive diagnosis of high grade glioma
* Patient whose surgery require the use of 5-ALA as standard of treatment

Exclusion Criteria:

* Patients who are not suitable for surgery
* Patients unable to provide informed consent due to cognitive impairment or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a presumptive diagnosis of high-grade glioma scheduled for surgical resection where 5-ALA is used as the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
5-ALA Fluorescence Detection Accuracy | Day of surgery (intra-operative ex-vivo analysis)
  Evaluation of the probe's sensitivity and specificity in detecting 5-ALA fluorescence signals in ex-vivo tumor tissue compared to the gold standard (histopathology/microscope). Measured parameters: operating wavelength interval, resolution, power range.

SECONDARY OUTCOMES:
Blood Vessel Identification | Day of surgery
  Ability of the probe (using ultrasound/Raman) to detect microvessels in the ex-vivo sample, correlated with histological microvessel density.
Tumor Cell Density Correlation | Day of surgery
  Correlation between the optical signal intensity and the tumor cell density assessed by pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Ciceri, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The Sponsor (Fondazione IRCCS Istituto Neurologico Carlo Besta) is the owner of the data resulting from the study. Dissemination of information or data requires the prior written consent of the Sponsor